CLINICAL TRIAL: NCT02552147
Title: Nicotinic Cholinergic Modulation as a Novel Treatment Strategy for Aggression Associated With Autism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1502015384
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Autism Spectrum Disorder; Aggression; Irritability
Keywords: Autism spectrum disorder; Aggression; Irritability; Nicotine; Nicotinic acetylcholine receptor; Nicotinic agonist; Adult autism
MeSH Terms: conditions — Autism Spectrum Disorder; Aggression; Autistic Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdermal nicotine first, placebo last (Experimental): Subject will receive transdermal nicotine 7 mg daily for 7 days, placebo patch for 7 days, then placebo patch for a final 7 days.
  Interventions: Drug: Transdermal nicotine; Other: Transdermal placebo
- Transdermal placebo first, nicotine last (Experimental): Subject will receive transdermal placebo daily for 7 days, placebo patch for another 7 days, then transdermal nicotine 7 mg daily for a final 7 days.
  Interventions: Drug: Transdermal nicotine; Other: Transdermal placebo

INTERVENTIONS:
Drug: Transdermal nicotine
Other: Transdermal placebo

SUMMARY:
Some individuals with autism spectrum disorders (ASD) also demonstrate irritability or aggression, which can interfere with functioning. The purpose of this pilot study is to test whether transdermal nicotine is effective for irritability and/or aggression in adults with ASD using a double-blind, placebo-controlled clinical trial. Subjects will participate in three visits. At the first visit, subjects are screened for eligibility and enrolled. Baseline measures include rating scales and a frustrative computerized task. They will then wear seven days of transdermal nicotine or placebo. Visit two is on day seven and the study measures are repeated, vital signs and side effects monitored. Subjects will return for a third and final visit on day 21 to repeat the study measures performed during visit two.

ELIGIBILITY:
Inclusion criteria:

* Age: 18-60
* Gender: All
* Language: Communicative in English
* Participants with a prior diagnosis of DSM-5 ASD at some point in their lifetime OR a DSM-4 diagnosis of Autism OR a DSM-4 diagnosis of Asperger's syndrome OR a DSM-4 diagnosis of Pervasive Developmental Disorder Not Otherwise Specified.
* Symptoms of irritability, agitation or aggression as reported by parent and/or participant
* Aberrant behavior checklist - Irritability Subscale (ABC-I) score of 16 or higher
* No changes in psychotropic medications within the past 14 days.
* Either lives with a primary caregiver or closely engaged with a primary caregiver who interacts with the patient daily
* BMI > 17.5 and < 45

Exclusion criteria:

* Age < 18 or > 60
* BMI < 17.5 or > 45
* Currently using tobacco or any nicotine products (transdermal, gum, e-cigarettes)
* Changes in psychotropic medication management within the past 14 days
* Previous allergy to transdermal patches
* Patients with heart rate > 100 or < 50 or known history of cardiac rhythm abnormalities
* Systolic blood pressure > 150 or < 95; diastolic blood pressure > 90 or < 50
* No symptoms of irritability, agitation, or aggression as reported by parent and/or participant
* ABC-I score of less than 16
* No primary caregiver, or primary caregiver unable to assist with rating scales

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09; Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Lewis, MD, PhD, Principal Investigator — Lecturer in psychiatry
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Placebo First, Nicotine Last: Subject will receive transdermal placebo daily for 7 days, placebo patch for another 7 days, then transdermal nicotine 7 mg daily for a final 7 days.
  Transdermal nicotine
  Transdermal placebo
- Transdermal Nicotine First, Placebo Last: Subject will receive transdermal nicotine 7 mg daily for 7 days, placebo patch for 7 days, then placebo patch for a final 7 days.
  Transdermal nicotine
  Transdermal placebo
Period: First Intervention (7 Days)
Arm/Group | Transdermal Placebo First, Nicotine Last | Transdermal Nicotine First, Placebo Last
Started | 4 | 4
Completed | 3 | 4
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Washout (7 Days)
Arm/Group | Transdermal Placebo First, Nicotine Last | Transdermal Nicotine First, Placebo Last
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Transdermal Placebo First, Nicotine Last | Transdermal Nicotine First, Placebo Last
Started | 3 | 4
Completed | 1 | 4
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: One subject was enrolled and randomized but later determined to be ineligible for the study and not included in the baseline analysis population.
Groups:
- All Study Participants: Participants randomized to receive either transdermal nicotine or placebo
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Aberrant Behavior Checklist-Irritability [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-irritability subscale measures irritability and related symptoms and the subscale score range is 0 (least symptomatic) to 45 (most symptomatic). The ABC is completed by parents/caregivers.
  units on a scale | 25 (8)
Aberrant Behavior Checklist-Lethargy/Social withdrawal [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-lethargy/social withdrawal subscale measures lethargy/social withdrawal and related symptoms and the subscale score range is 0 (least symptomatic) to 48 (most symptomatic). The ABC is completed by parents/caregivers.
  units on a scale | 20 (13)
Aberrant Behavior Checklist-Stereotypic behavior [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-stereotypic behavior subscale measures stereotypic behaviors and related symptoms and the subscale score range is 0 (least symptomatic) to 21 (most symptomatic). The ABC is completed by parents/caregivers.
  units on a scale | 9 (7)
Aberrant Behavior Checklist-Hyperactivity [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-hyperactivity subscale measures hyperactivity and related symptoms and the subscale score range is 0 (least symptomatic) to 48 (most symptomatic). The ABC is completed by parents/caregivers.
  units on a scale | 26 (11)
Aberrant Behavior Checklist-Inappropriate speech [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-Inappropriate speech subscale measures Inappropriate speech and related symptoms and the subscale score range is 0 (least symptomatic) to 12 (most symptomatic). The ABC is completed by parents/caregivers.
  units on a scale | 6 (4)
Social Responsiveness Scale-2 [Mean (Standard Deviation); unit: units on a scale] — The Social Responsiveness Scale (SRS) - 2 quantifies impairments in social behaviors seen in autism spectrum disorder and related conditions and their severity. The version used in this study is completed by parents/caregivers. The raw score range is 0 (unaffected) to > 134 (extremely affected). The ABC is completed by parents/caregivers.
  units on a scale | 177 (25)
Number on antipsychotic medication [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Aberrant Behavior Checklist Irritability Subscale (ABC-I)
Description: Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-irritability subscale measures irritability and related symptoms and the subscale score range is 0 (least symptomatic) to 45 (most symptomatic). The ABC is completed by parents/caregivers.
Time Frame: Baseline and 7 days.
Population: All participants who completing all study visits and for which ratings scales were completed in accordance with study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nicotine: Subject receiving transdermal nicotine in either the first or last week of the study and completing all study visits.
- Placebo: Subject receiving transdermal placebo in either the first or last week of the study and completing all study visits.
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -12 (3) | -7 (8)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .44, Wilcoxon (Mann-Whitney); Two-tailed

2. Secondary Outcome: Change in Social Responsiveness Scale-Adults (SRS-A)
Description: The Social Responsiveness Scale (SRS) - 2 quantifies impairments in social behaviors seen in autism spectrum disorder and related conditions and their severity. The version used in this study is completed by parents/caregivers. The raw score range is 0 (unaffected) to > 134 (extremely affected). The ABC is completed by parents/caregivers.
Time Frame: Baseline and 7 days.
Population: All participants completing all study visits and for which ratings scales were completed in accordance with study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -1 (25) | -15 (23)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney); Two-tailed

3. Secondary Outcome: Change in Qualitative Description of Irritability and Aggression Symptoms
Description: Brief qualitative reports of the patient's subjective experience will be recorded by asking "In what ways did you find the patch helpful or harmful during the past week, if at all?".
Time Frame: Baseline and 7 days
Population: Data were not collected.
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Frustration and Irritability Ratings During Frustration-induction Go-NoGo Task
Description: Subjects will perform a computerized frustration-induction task and complete a rating scale of irritability and frustration levels.
Time Frame: Baseline and one week
Population: Data were not collected.
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in State/Trait Anxiety Inventory (STAI) Score
Description: The State-Trait Anxiety Inventory (STAI) is a measure of trait and state anxiety. It ranges from a score of 20 (least affected) to 80 (most affected).
Time Frame: Baseline and day 7
Population: Data were not collected.
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Nightly Sleep Quality
Description: Caregivers rated nightly sleep quality from 0 (worst) to 10 (best). Average rating for each treatment week is compared.
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 10 (0.2) | 9 (2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney); Two-tailed

7. Post Hoc Outcome: Aberrant Behavior Checklist - Lethargy/Social Withdrawal Subscale Change From Baseline
Description: Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-lethargy/social withdrawal subscale measures lethargy/social withdrawal and related symptoms and the subscale score range is 0 (least symptomatic) to 48 (most symptomatic). The ABC is completed by parents/caregivers.
Time Frame: Baseline and 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -2 (3) | -7 (4)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney); Two-tailed

8. Post Hoc Outcome: Aberrant Behavior Checklist - Stereotypic Behavior Subscale Change From Baseline
Description: Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-stereotypic behavior subscale measures stereotypic behaviors and related symptoms and the subscale score range is 0 (least symptomatic) to 21 (most symptomatic). The ABC is completed by parents/caregivers.
Time Frame: Baseline and 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -2 (3) | -4 (4)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney); Two-tailed

9. Post Hoc Outcome: Aberrant Behavior Checklist - Hyperactivity Subscale Change From Baseline
Description: Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-hyperactivity subscale measures hyperactivity and related symptoms and the subscale score range is 0 (least symptomatic) to 48 (most symptomatic). The ABC is completed by parents/caregivers.
Time Frame: Baseline and 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -7 (6) | -6 (6)
Statistical Analysis 1: Comparison: Nicotine vs Placebo; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney) — P value was calculated to >0.99 and thus rounded to 1.0; Two-tailed

10. Post Hoc Outcome: Aberrant Behavior Checklist - Inappropriate Speech Subscale Change From Baseline
Description: Aberrant Behavior Checklist (ABC) measures symptom subscales for individuals with neurodevelopmental disorders. The ABC-Inappropriate speech subscale measures Inappropriate speech and related symptoms and the subscale score range is 0 (least symptomatic) to 12 (most symptomatic). The ABC is completed by parents/caregivers.
Time Frame: Baseline and 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -1 (2) | 0.2 (0.8)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney); Two-tailed

11. Post Hoc Outcome: Global Aggressive Behavior Improvement
Description: Caregivers asked which treatment week showed the greatest improvement in aggressive or irritable behavior
Time Frame: Baseline and 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 4 | 2
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.69, Binomial test

ADVERSE EVENTS:
Time Frame: Duration of trial (3 weeks).
Arm/Group | Nicotine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine (N=7) | Placebo (N=7)
Nightmare (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Unable to recruit the pre-specified number of subjects; Subjects were unable to reliably complete personal ratings (STAI and STAXI) and were unable to reliably complete the frustrative computer task.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT02552147/Prot_SAP_002.pdf
  • Informed Consent Form (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT02552147/ICF_001.pdf